CLINICAL TRIAL: NCT02868424
Title: Early Phase I Study of the Safety and Preliminary Efficacy of Human Fetal Retinal Pigment Epithelial(fRPE) Cells Subretinal Transplantation in Age-Related Macular Degeneration(AMD) Patients
Brief Title: Treatment of Age-related Macular Degeneration by Fetal Retinal Pigment Epithelial Cells Transplantation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-fRPE-001
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Age Related Macular Degeneration; Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fRPE cells (Experimental): Subretinal transplantation of fRPE cells in experimental eye
  Interventions: Drug: fRPE cells

INTERVENTIONS:
Drug: fRPE cells — fRPE cells transplantation directly into the subretinal space of one eye (experimental eye) in a single transplant procedure
  Other Names: human fetal retinal pigment epithelial cells

SUMMARY:
Early Phase I Study of the Safety and Preliminary Efficacy of Human Fetal Retinal Pigment Epithelial(fRPE) Cells Subretinal Transplantation in Age-Related Macular Degeneration(AMD) Patients

DETAILED DESCRIPTION:
This study is a perspective, single-arm and open-labeled investigation of the safety and preliminary efficacy of unilateral subretinal transplantation of fRPE cells in subjects with dry Age-Related Macular Degeneration and non-exudative AMD. The investigators will recruit and enroll 6 patients based on specific inclusive/exclusive criteria. Experimental and self-controlled eye will be determined based on best-corrected visual acuity (BCVA). The eye with BCVA of no more than 20/400 will be determined as experimental eye, which will be divided into 3 groups and undergo subretinal injection of 3 different dosages of fRPE cells (100.000, 200,000 or 500,000) respectively, while the other one (BCVA of more than or equal to 20/400) as control eye, will not receive the surgery.

fRPE cells will be obtained from the fetuses aborted in the Department of Obstetrics and Gynecology in Jiangsu Province Hospital from 2015 to 2018. The obtained fRPE cells will meet specific inclusive/exclusive criteria and conform to Good manufacturing practices (GMP). fRPE will be transplanted by a board-certified vitreoretinal surgeon, which will be administered into the subretinal space of experimental eye through a standard surgical approach.

Immunosuppressive agents will be administered orally to all subjects after transplantation. Dosage and time duration of immunosuppressive agents will be regulated strictly relying on the condition of immune rejection. Subjects will be monitored with ophthalmologic and systemic examinations frequently at regular post-transplant intervals after fRPE cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dry AMD or non-exudative AMD (geographical atrophy>250μm, involving central fovea of macular; or AMD with fibrous disciform scar and maintained stationary for at least 3 months)
* Experimental eye with best-corrected visual acuity (BCVA) of no more than 20/400 and control eye with BCVA of more than or equal to 20/400
* Patients are in good state
* Patient understand and sign the consent form.

Exclusion Criteria:

* Blood routine examination is abnormal (hemoglobin<10gm/dL; blood platelet count<100k/mm³; neutrophil count<1000/mm³)
* Blood biochemistry is abnormal (ALT／AST>1.5; creatinine>1.3mg/dL)
* Experimental eye has optic nerve atrophy caused by glaucoma
* Patients need cataract surgery within a year
* Patients have received cataract surgery and other ocular surgery in recent 3 months
* Experimental eye has retinal detachment, or has received retinal detachment surgery.
* Patients with uveitis and other endophthalmitis
* Patients with other ocular disease affecting vision.
* Patients have participated in clinical study of ocular or systemic drug use in recent 6 months.
* Patients with medical history of malignant cancer (except resected basal cell carcinoma and squamous-cell carcinoma).
* Patients with medical history of myocardial infarction
* Patient with diabetes
* Patient with Parkinson disease or Alzheimer's disease
* Patients are under the treatment of immunosuppressive agent (except intermittent, low-dose corticosteroid treatment).
* Patients with other medical conditions that restricts the compliance and safety of patients, or affects experimental results.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-13 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Two years following transplantation
  Descriptive analysis of frequency and types of adverse events experienced by each subject during the study period.

SECONDARY OUTCOMES:
Assessment of standardized ETDRS acuity testing | Two years following transplantation
  ETDRS stands for Early Treatment Diabetic Retinopathy Study which is designed to accurately measure visual acuity via ETDRS Scoring.
Assessment of visual function changes | Two years following transplantation
  Assessments will include fluorescein angiography, fundus photography, spectral domain ocular coherence tomography (SD-OCT), microperimetry and multifocal electroretinography.
Assessment of systemic condition | Two years following transplantation
  Items will include vital signs, electrocardiogram, blood and urine routine examination, tumor marker.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghuai Liu, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes